CLINICAL TRIAL: NCT01387087
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of ASP015K Following Single Oral Doses to Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP015K
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Clinical Trials Registry, Astellas Pharma Global Developmnt
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: 015K-CL-HV01
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP015K
Keywords: ASP015K; Healthy subjects; Pharmacodynamics; Maximum tolerated dose
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- Group A (Experimental): Lowest dose, all males, fasting
  Interventions: Drug: ASP015K
- Group B (Experimental): Second lowest dose, all males, fasting
  Interventions: Drug: ASP015K
- Group C (Experimental): Third lowest dose, all males, fasting
  Interventions: Drug: ASP015K
- Group D (Experimental): Middle dose, all males, fasting
  Interventions: Drug: ASP015K
- Group E (Experimental): Third lowest dose, all females, fasting
  Interventions: Drug: ASP015K
- Group F (Experimental): Third highest dose, all males, fasting then fed
  Interventions: Drug: ASP015K
- Group G (Experimental): Second highest dose, all males, fasting
  Interventions: Drug: ASP015K
- Group H (Experimental): Highest dose, all males, fasting
  Interventions: Drug: ASP015K
- Group I (Experimental): Second highest dose, all females, fasting
  Interventions: Drug: ASP015K
- Placebo Group A (Placebo Comparator): all male, fasting
  Interventions: Drug: Placebo
- Placebo Group B (Placebo Comparator): all male, fasting then fed
  Interventions: Drug: Placebo
- Placebo Group C (Placebo Comparator): all female, fasting
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP015K — oral
  Arms: Group A; Group B; Group C; Group D; Group E; Group F; Group G; Group H; Group I
Drug: Placebo — oral
  Arms: Placebo Group A; Placebo Group B; Placebo Group C

SUMMARY:
The objective of the study is to explore safety and tolerability of single ascending doses of ASP015K, establish the maximum tolerated dose, and determine the pharmacokinetics and pharmacodynamics in healthy volunteers.

DETAILED DESCRIPTION:
Subjects will be confined to the clinical research unit for five days. Some subjects will participate in two confinement periods. Subjects will receive a follow-up phone call to assess safety seven days after the administration of the single dose of study drug.

Subjects will be assigned to one of nine sequential groups A, B, C, D, E, F, G, H, or I. In each group, 6 subjects will be randomized to ASP015K and 2 subjects will be randomized to placebo. Subjects in group F will participate in two treatment periods. Subjects in the first treatment period of group F will have a single study drug dose administered in the fasted state. Subjects in the second treatment period of group F will have a single study drug dose administered immediately following a standard FDA recommended high-fat breakfast.

ELIGIBILITY:
Inclusion Criteria:

* If female, the subject is at least 2 years post menopausal or is surgically sterile per documentation provided by a third party medical professional and the subject is not pregnant as documented by a negative serum pregnancy test
* If male, the subject agrees to sexual abstinence and/or to use a highly effective method of birth control during the study period
* Subject is medically healthy, with no clinically significant abnormalities on medical history or abnormalities observed upon physical examination or 12 lead electrocardiogram (ECG)
* Subject's fasting clinical laboratory values are within normal limits
* Subject is a non-smoker and has not used tobacco for a minimum of 3 months
* Subjects must weigh at least 45 kg and have a Body Mass Index (BMI) of 18-32 kg/m2

Exclusion Criteria:

* Subject has a positive test for hepatitis C antibody, or positive for hepatitis B surface antigen (HBsAg)
* Subject has a history of the human immunodeficiency virus (HIV) antibody
* Subject has a history of severe allergic or anaphylactic reactions
* Subject has a history of chronic diarrhea
* Subject has been vaccinated within the last 60 days prior to study drug administration
* Subject has a previous history of any clinically significant neurological, gastrointestinal, renal, hepatic, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, or any other medical condition that, in the Investigator's opinion, would preclude participation in the study
* Subject has had clinically significant illness within 1 month prior to study drug administration
* Subject has a history of hemorrhoids
* Subject has a history of drug or alcohol abuse or a positive urine screen for alcohol or drugs of abuse and/or illegal drugs
* Subject has had treatment with prescription medication (except hormone replacement therapy and acetaminophen), complementary and alternative medicines (CAM) within 14 days, over-the-counter products within 1 week, or alcohol, caffeine or grapefruit juice within 24 hours prior to study drug administration
* Subject has had treatment with another investigational drug or approved therapy for investigational use within 30 days or 10 half-lives, whichever is longer, prior to study drug administration or has participated in a prior group in the current study
* Subject has a history of blood donation within 30 days prior to study drug administration or has donated plasma within 7 days prior to study drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed through vital signs, electrocardiograms (ECGs), physical exams, reports of adverse events, and analysis of blood and urine samples | 8 days
Pharmacokinetic assessment through the analysis of blood and urine samples | Up to Day 4
Pharmacodynamic assessment through the analysis of blood samples | Up to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Prism Research, Saint Paul, Minnesota